CLINICAL TRIAL: NCT05550285
Title: Patient Specific 3D Printed Titanium Mesh Versus Computer Guided Calvarial Bone Graft for Orbital Floor Reconstruction: A Randomized Clinical Trial
Brief Title: 3D Printed Titanium Mesh vs Guided Autogenous Graft
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mohammed Ghassan Mohammed Shaalan (Other)
Responsible Party: Sponsor-Investigator, Mohammed Ghassan Mohammed Shaalan, Master Student, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMFS 3-3-10
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Orbital Floor (Blow-Out) Open Fracture; Enophthalmos Traumatic
Keywords: Blow-out Fracture, Orbital floor Fracture , Orbital Floor Reconstruction
MeSH Terms: conditions — Fractures, Open; Orbital Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Orbital Volume After Using Guided Calvarial Graft in Floor Recontsruction (Experimental)
  Interventions: Device: orbital floor recontriction
- Orbital Volume After Using 3D Printed Titanium mesh in Floor Recontsruction (Experimental)
  Interventions: Device: orbital floor recontriction

INTERVENTIONS:
Device: orbital floor recontriction — Guided Calvarial Graft Harvesting vs 3D Printed Titanium mesh

SUMMARY:
In this study, the hypothesis states that there is no significant difference between specified populations. In our case, the 3D printed patient-specific titanium mesh is thought to have the same effect and results in comparison with the computer-guided calvarial bone graft technique according to the related studies.

DETAILED DESCRIPTION:
Recruitment:

Patients' data will be enrolled in the database of the Outpatient clinics of the Department of Oral & Maxillofacial Surgery, Faculty of Dentistry, Cairo University

* If there is potential eligibility, the patient will be examined thoroughly as described before.
* Consecutive sampling is done through screening of patients. This will continue until the target population is achieved.
* Identifying and recruiting potential subjects is achieved through a patient database

Pre-operative data Collection:

All Patients will undergo CT scan and throughout medical history will be taken. Enophthalmos and orbital volume will be measured via CT data using DICOM viewers, the anterior orbital boundary is defined by a line joining the zygomatico-frontal process on each side. Cross-sectional area is measured using the region of interest (ROI) facility, after tracing the orbital outline The degree of enophthalmos is assessed by measuring the distance between the posterior surface of each lens and the anterior orbital boundary line.

Exophthalmometer The instrument is placed on the lateral orbital rim of each side, using as small of a base as possible, the device measures the distance between the lateral orbital rim and the most anterior position of the cornea.

For Both Groups, the retrieved DICOM files of the CT scan will be imported in a DICOM (Digital Imaging and Communications in Medicine) viewer software (Mimics 19.0; Mimics Medical 19.0, Materialise, Leuven, Belgium) and segmentation will be done starting from thresholding and region growing to form a mask for the area of interest.

For Control Group, the orbital defect outline will be identified and measured and the same measurements will be transferred to the parietal bones bilaterally taking into consideration that they must be in the thickest portion of the parietal bone to construct the surgical guide prior to surgery. A three-dimensional model of the patient's skull will be calculated from the selected mask; the skull model will be manufactured and printed and will be used to assure seating of the Autogenous graft intra-operatively before inserting it in the surgical field.

For Study Group, the orbital floor defect will be digitally reconstructed by mirroring an individually defined 3-dimensional (3D) segment from the unaffected side onto the deformed side to determine the locations and range of orbital defects. The Standard Template Library data transformed from the 3D data will be used in the creation computer-assisted 3D Printed titanium mesh implant. The implants will be designed based on the PorousiTi structure which was created to replicate the mechanical properties of human bone. Anatomical obstacles including infra-orbital nerve and lacrimal duct were taken into account during this process.

Intra operative procedures for both groups: A vasoconstrictor will be injected under the conjunctiva to aid in hemostasis, Additional solution will be infiltrated during the lateral canthotomy. A corneal shield will be placed to protect the globe and the lower eyelid will be everted with fine forceps and two or three traction sutures will be placed through the eyelid. These sutures will be placed straight through the eyelid, from palpebral conjunctiva to skin, approximately 4 to 5 mm below the eyelid margin to ensure that the tarsal plate is included in the suture.

When a lateral canthotomy is indicated, the canthotomy will be the initial incision. One tip of the pointed scissors is inserted within the palpebral fissure, extending laterally to the depth of the underlying lateral orbital rim (approximately 7 to 10 mm). The scissors are used to cut horizontally through the lateral palpebral fissure. The structures that are cut in the horizontal plane are the skin, orbicularis oculi muscle, orbital septum, lateral canthal tendon, and conjunctiva.

The traction sutures are used to evert the lower eyelid. The lower eyelid is still tethered to the lateral orbital rim by the inferior limb of the lateral canthal tendon. The tendon, which is easily visualized with eyelid retraction, will be released with a sharp vertical cut. When performing the cantholysis, the scissors must be positioned with a vertical orientation. After cantholysis, the lower eyelid will be immediately freed from the lateral orbital rim, making the eversion more effective.

After the lower eyelid is everted, the position of the lower tarsal plate through the conjunctiva will be noted. Incising in the conjunctiva, blunt-tipped pointed scissors are used to dissect through the small incision in the conjunctiva made during the lateral canthotomy, inferiorly toward the infraorbital rim. Traction sutures are used to evert the lower eyelid during the dissection. The scissors are spread to clear a pocket posterior to the orbital septum, ending just posterior to the orbital rim Scissors are used to incise the conjunctiva and lower eyelid retractors midway between the inferior margin of the tarsal plate and the inferior conjunctival fornix. The incision can be extended as far medially as necessary for the surgery but must not violate the lacrimal sac.

The incised edge of the vestibular conjunctiva can be dissected free, providing a location for a traction suture to hold the corneal shield in place.

After retracting the orbital contents internally and the lower eyelid externally, using suitable retractors, the periorbita will be sharply incised, avoiding the lacrimal sac medially. During the retroseptal approach, the incision through the periorbita is immediately posterior to the orbital rim. Periosteal elevators are used to strip the periosteum over the orbital rim and anterior surface of the maxilla and zygoma, and the orbital floor. A broad malleable retractor should be placed as soon as feasible to protect the orbit and to confine any herniating periorbital fat.

For Study group: After identification of the floor defect, Patient-Specific titanium mesh that will be manufactured and printed by CAD-CAM technology to cover the defect and will be seated by the operator and assure that there is no entrapment of tissue underneath the mesh.

In Control group: In preparation of the patient, hair may or may not be shaved, depending on the clinical situation.

If exposure of zygomatic arch, orbital rim or temporomandibular joint will be also needed, a coronal incision will be designed, the coronal flaps may be retracted to expose the parietal region. A vasoconstrictor will be injected into the subgaleal plane to promote hemostasis and to help separate the tissue layers. Another technique for hemostasis involves inserting running blocking sutures of 2-0 polypropylene or nylon along each side of the proposed incision line. These sutures will be removed at the completion of scalp closure. the last technique, special cautery scalpels are used for scalp incisions, but these heated scalpels may damage hair follicles.

Otherwise, a laterally placed incision in the parieto-temporal region is used. If possible, the incision should be designed away from the graft site, as there is a tendency for the incision to scar down to the underlying graft bed.

The surgical guide will be positioned and checked for stability and accuracy. The borders of the required graft will be marked using a micro-disk, and then the osteotomy will be further deepened to the spongy diploe of the skull bone. Once the required level is reached, undermining will be performed with bone chisels until the outer table of the bone lock is freed, then the bone block will be inserted and seated on the Printed Skull Model to assure stability and then inserted on orbital floor to cover the defect and prevent any entrapment of orbital fibrous-adipose-muscular tissues. The surgical field will be rinsed with saline and then closed by absorbable sutures, followed by cutaneous needles stapled to the skin of the scalp.

In both groups:

Forced duction test will be repeated to rule out iatrogenic entrapment, and the position of the orbital floor implant will be once again checked to ensure that no migration had occurred during the forced duction testing.

Inferior canthopexy suture will be inserted but not tied, the conjunctiva then sutured, a 4-0 polyglactin or other long-lasting suture is used to reattach the lateral portion of the inferior tarsal plate to the residual superior portion of the lateral canthal tendon or to the fixed surrounding tissues.

The suture through the lateral border of the lower tarsus and/or cut portion of the lateral canthal tendon may be facilitated by elevating the skin sharply with a blade No 15, slightly atop the canthus or tarsal plate. The conjunctiva should be closed with a running 6-0 chromic gut suture. The ends of the suture may be buried. The inferior canthopexy suture is then tightened and tied, drawing the lower eyelid into position. Finally, subcutaneous sutures and 6-0 skin sutures are placed along the horizontal lateral canthotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous fresh maxillofacial trauma within 14 days affecting zygomatic bones and orbital walls.
* Patients with medical history that did not hinder previous reconstruction of orbital floor defect.
* Both genders males and females will be included.

Exclusion Criteria:

* Patients with craniofacial anomalies or syndromes.
* Subjected to irradiation in the head and neck area less than 6 months to -1 year before procedure
* Pregnant or nursing females.
* Psychiatric problems or unrealistic expectations.
* Immunosuppressed or immunocompromised patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Orbital volume Measuring | Immediately Post Operative

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Farid Shehab, Professor, Study Director — Professor, Oral & Maxillofacial surgery, Cairo University; Heba Mohamed Kamel, Assistant Professor, Study Director — Assistant professor, Oral & Maxillofacial surgery, Cairo University
Locations (1):
- Mohammed Ghassan Mohammed Shaalan, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided